CLINICAL TRIAL: NCT01773291
Title: Adjuvant Acupuncture Therapy in Patients With Severe Head Injury: a Randomized Controlled Trial
Brief Title: Adjuvant Acupuncture for Severe Head Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMRPG8B1211; 103-5150C (Other: Chang Gung Medical Foundation Institutional Review Board)
Record Dates: First submitted 2013-01-11; First posted 2013-01-23 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-07

CONDITIONS: Head Injury
Keywords: Acupuncture; laser acupuncture; traumatic brain injury
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- acupuncture (Experimental): acupuncture on GV26 and 12 Well points
  Interventions: Other: acupuncture
- laser acupuncture (Experimental): laser acupuncture on GV26 and 12 Well points
  Interventions: Other: laser acupuncture
- control group (Sham Comparator): laser acupuncture without laser output in control group.
  Interventions: Other: control

INTERVENTIONS:
Other: acupuncture — acupuncture on GV26 and 12 Well points
  Arms: acupuncture
Other: laser acupuncture — laser acupuncture on GV26 and 12 Well points
  Arms: laser acupuncture
Other: control — sham laser acupuncture
  Arms: control group

SUMMARY:
The purpose of this study is to determine the therapeutic effect of acupuncture on severe head injury under conventional treatment. A double-blind clinical trial is conducted up to 6 weeks and the change of subjects' Glasgow coma scale (GCS) and muscle power is measured.

DETAILED DESCRIPTION:
Objective: To investigate the therapeutic effect of acupuncture on severe head injury under conventional treatment.

Methods: 90 subjects aged 12 to 70 years with severe head injury (Glasgow coma scale score 8 or less) are randomly divided into acupuncture, laser acupuncture and control group. We use restoring consciousness acupuncture (GV26 and 12 Well points) to treat the subjects 3 sessions per week under conventional treatment at Department of Neurosurgery. A double-blind clinical trial is conducted up to 6 weeks and the change of subjects' GCS and muscle power is measured.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 12 to 70 years with severe head injury (Glasgow coma scale score 8 or less)
* with informed consent

Exclusion Criteria:

* dilated pupils without light reflex
* serious complications during therapeutic course
* interruption of therapeutic course
* unfavored condition assessed by physician in charge
* without informed consent

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Long Hu, MS, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] DeFina PA, Fellus J, Thompson JW, Eller M, Moser RS, Frisina PG, Schatz P, Deluca J, Zigarelli-McNish M, Prestigiacomo CJ. Improving outcomes of severe disorders of consciousness. Restor Neurol Neurosci. 2010;28(6):769-80. doi: 10.3233/RNN-2010-0548. PMID 21209492
- [Background] Jennett B, Adams JH, Murray LS, Graham DI. Neuropathology in vegetative and severely disabled patients after head injury. Neurology. 2001 Feb 27;56(4):486-90. doi: 10.1212/wnl.56.4.486. PMID 11222792
- [Result] Clauss R, Nel W. Drug induced arousal from the permanent vegetative state. NeuroRehabilitation. 2006;21(1):23-8. PMID 16720934
- See also: Acupuncture for Disorders of Consciousness - A Case Series and Review — http://www.intechopen.com/books/acupuncture-clinical-practice-particular-techniques-and-special-issues/acupuncture-for-disorders-of-consciousness-a-case-series-and-review
- See also: Efficacy of Stimulation at the Jing-Well Points of Meridians — http://dx.doi.org/10.15344/2394-4978/2015/121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with severe traumatic brain injury (Glasgow Coma Scale, GCS ≤ 8) admitted to neurosurgical intensive care unit (NSICU) were enrolled and randomly divided into three groups sequentially.
Pre-assignment Details: Exclusion criteria: dilated pupils without light reflex, unstable vital signs, serious complication during therapeutic course, serious multiple injuries, withdrawal by subject, physician decision, without informed consent.
Groups:
- Acupuncture: acupuncture on Shuigou (GV26) and 12 Well points
  acupuncture: acupuncture on GV26 and 12 Well points
- Control Group: laser acupuncture without laser output in control group.
  control: sham laser acupuncture on GV26 and 12 Well points
Period: Overall Study
Arm/Group | Acupuncture | Laser Acupuncture | Control Group
Started | 8 | 9 | 7
Completed | 7 | 9 | 6
Not Completed | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Laser Acupuncture | Control Group | Total
Number analyzed (Participants) | 7 | 9 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.29 (17.14) | 49.11 (16.86) | 47.17 (21.47) | 45.77 (17.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 6 | 7 | 4 | 17
Region of Enrollment [Number; unit: participants]
  Taiwan | 7 | 9 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Glasgow Coma Scale (GCS)
Description: Eye response (E)
  There are four grades starting with the most severe:
  1. No eye opening
  2. Eye opening in response to pain stimulus.
  3. Eye opening to speech.
  4. Eyes opening spontaneously Verbal response (V)
  There are five grades starting with the most severe:
  1. No verbal response
  2. Incomprehensible sounds.
  3. Inappropriate words.
  4. Confused.
  5. Oriented. Motor response (M)
  There are six grades:
  1. No motor response
  2. Decerebrate posturing accentuated by pain
  3. Decorticate posturing accentuated by pain
  4. Withdrawal from pain
  5. Localizes to pain
  6. Obeys commands
  The sum of the score was measured (3 - 15) before and after treatment during hospitalization. The higher score, the better outcome.
Time Frame: 6 weeks
Population: The subjects were treated 3 times a week (maximum 18 sessions in 6 weeks). The GCS was measured before and after treatment during hospitalization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Laser Acupuncture | Control Group
Number analyzed (Participants) | 7 | 9 | 6
units on a scale | 3.14 (1.46) | 3.11 (3.02) | 4.67 (2.73)

2. Secondary Outcome: Muscle Power (MP)
Description: Medical Research Council (MRC) muscle-grading scale Grade MRC grade of muscle strength 0 No movement
  1. Flicker of movement only
  2. Movement possible when assisted by gravity or gravity is eliminated
  3. Movement possible against gravity but without imposed resistance
  4. Weak movement possible against gravity
  5. Normal movement against gravity and against imposed resistance
  The 4 muscle groups were assessed on the 0 to 5 scale and scores were summed before and after treatment during hospitalization. The total score ranges from 0-20, with higher score indicating better outcome.
Time Frame: 6 weeks
Population: The subjects were treated 3 times a week (maximum 18 sessions in 6 weeks). The MP was measured before and after treatment during hospitalization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Laser Acupuncture | Control Group
Number analyzed (Participants) | 7 | 9 | 6
units on a scale | 4.29 (4.46) | 4.33 (3.39) | 2.83 (3.49)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Acupuncture | Laser Acupuncture | Control Group
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 0/6

LIMITATIONS AND CAVEATS:
Inclusion criteria leading to small numbers (24/583 in 2.5 years) of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes